CLINICAL TRIAL: NCT03632187
Title: To Demonstrate the Ability of Abatacept in Comparison to Placebo to Obtain a Low Disease Activity [PMR-AS (CRP) Lower or Equal to 10] Without GCs (Prednisone or Prednisolone) at Week 12 in Early Onset PMR Patients.
Brief Title: Abatacept in earLy Onset Polymyalgia Rheumatica: Study ALORS
Acronym: ALORS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Brest (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 29BRC17.0228 _ALORS
Record Dates: First submitted 2018-07-11; First posted 2018-08-15 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Polymyalgia Rheumatica
MeSH Terms: conditions — Polymyalgia Rheumatica | interventions — Abatacept

STUDY DESIGN:
Intervention Model Description: This is a multicenter double blinded randomized placebo controlled trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Subcutaneous abatacept every weeks during 3 months (W0 to W11). Then, at W12, if PMR-AS>10, they will receive GCs according to the PMR-AS (PMR-AS≤10: no GCs, PMR-AS between 10-20: 10mg/day, PMR-AS between 21-30: GCs at 15mg/d and if PMR-AS> 30: 20mg/d). Dosage of GCs will be decreased between W16 and W24 (1mg every week) in each arm according to PMR-AS (PMR-AS < 10: decrease, PMR-AS > 17 increase to previous dosage, 10 ≤ PMR-AS ≤ 17: stable dose). If PMR-AS ≤10, the patients wont receive any treatment until a flare.
  Interventions: Drug: Abatacept
- Control group (Placebo Comparator): Subcutaneous placebo every week during 3 months (W0 to W11). Then, at week 12, if PMR-AS>10, they will receive GCs according to the PMR-AS (PMR-AS≤10: no GCs, PMR-AS between 10-20: 10mg/day, PMR-AS between 21-30: GCs at 15mg/d and if PMR-AS> 30: 20mg/d). Dosage of GCs will be decreased between W16 and W24 (1mg every week) in each arm according to PMR-AS (PMR-AS < 10: decrease, PMR-AS > 17 increase to previous dosage, 10 ≤ PMR-AS ≤ 17: stable dose). If PMR-AS ≤10, the patients won't receive any treatment until a flare.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Abatacept — Subcutaneous abatacept every weeks during 3 months
  Arms: Experimental group
Drug: Placebos — Subcutaneous placebo every week during 3 months
  Arms: Control group

SUMMARY:
Polymyalgia rheumatic (PMR) is a frequent inflammatory disease. It affects the elderly, with peak incidences at the age of 70 to 80 years; an age >50 years or older, is considered a criterion for the diagnosis. Polymyalgia rheumatica occurs at a frequency that is 3 to 10 times that of giant-cell arteritis. Disease risk varies according to race and geographic region. The incidence is highest among whites in northern European populations (about 20 cases per 100,000 persons older than 50 years of age); it is lower in southern European populations (about 10 cases per 100,000).The diagnosis is based on established ACR/EULAR classification criteria.

Long term low-dose glucocorticoid (GCs) (prednisone or prednisolone started at 15 to 20 mg/day progressively tapered) is the mainstay of the treatment.

The activity of PMR is evaluated using the PMR-AS, a disease activity score based on morning stiffness, ability to elevate the upper limbs, physician's global disease assessment and pain assessment measured by the patient using VAS, and the C-reactive protein (CRP) level. The PMR-AS is considered as relevant to define relapse and remission but also to decide if treatment have to be decreased, unchanged or increased (PMR-AS < 10: decrease, PMR-AS > 17 increase to previous dosage, 10 ≤ PMR-AS ≤ 17: stable dose)..

Comorbidity in PMR are due to GCs and 30% of the patients underwent a relapse when tapering GCs. If the investigators able to start prednisone at a lower dosage (i.e. 8 mg then tapered for 3 to 4 months), the cumulative dosage of steroid would not have major side effects but it is not possible without new therapeutic agents.

The TENOR study (Tolerance and Efficacy of tocilizumab iN pOlymyalgia Rheumatica), a phase 2 study, demonstrated efficacy of tocilizumab as first line treatment in PMR without GCs and its ability to spare GCs. This was the first study demonstrating that a biologic may improve PMR without steroid, and that also showed that a short treatment by biologic followed by a low dose GCs therapy may be a new concept in the treatment of PMR.

Molecular studies in GCA and PMR suggest that dendritic cells initiate the pathogenic cascade and recruit T cells. Two major immune-response networks have been identified related to type 1 helper T-cell (Th1) and to helper T-cell (Th17). Abatacept is comprised of the ligand-binding domain of CTLA4 plus modified Fc domain derived from IgG1. By containing CTLA4, abatacept blocks the engagement of CD28 with its ligand, thereby inhibiting T cell activation. It has recently demonstrated its efficacy in Granulomatosis with polyangiitis (GPA) but also in giant cell arteritis (GCA). Due to its good safety profile in rheumatoid arthritis and its potential to modulate T cell activation and derived cytokines, abatacept is an attractive agent to investigate in patients with PMR.

In this randomized prospective placebo controlled study, the objective is to demonstrate the ability of abatacept to improve alone PMR and then to allow a steroid sparing effect after this induction treatment, in early onset PMR.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 50 years
* Fulfilling ACR/EULAR criteria
* Disease duration≤6 months
* No steroid since 2 weeks prior randomization
* PMR-AS≥ 17
* Absence of signs or symptoms of other musculoskeletal or connective tissue conditions
* Able to give informed consent
* Concomitant treatments with methotrexate or hydroxychloroquine are not permitted.

Exclusion Criteria:

* Clinical symptoms of giant cell arteritis
* Uncontrolled high blood pressure or cardiovascular disease
* Clinical evidence of significant unstable or uncontrolled acute or chronic diseases not due to PMR
* Planned surgical procedure or medical history, blood abnormalities or any clinical condition that compromises inclusion
* History of malignant neoplasm within the last 5 years.
* Current active infection not controlled
* Detailed exclusion criteria related to prior or concomitant therapy, general safety and laboratory data are reported in the protocol

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2022-07-21 (Estimated)

PRIMARY OUTCOMES:
Following of one biological parameter (CRP) | 12 weeks
  The Polymyalgia Rheumatica Activity score is evaluated with a biological parameter named CRP.

SECONDARY OUTCOMES:
Emergence of adverse events (Safety and tolerability) | 36 weeks
  The safety is evaluated with the adverse events in both arms
Following of the Polymyalgia Rheumatica Activity score | 36 weeks
  The Polymyalgia Rheumatica Activity score is evalauted with CRP and without CRP. The activity of Polymyalgia Rheumatica is evaluated using the Polymyalgia Rheumatica Activity score (PMR-AS), a disease activity score based on morning stiffness, ability to elevate the upper limbs, physician's global disease assessment and pain assessment measured by the patient using VAS, and the C-reactive protein (CRP) level. The PMR-AS is considered as relevant to define relapse and remission but also to decide if treatment have to be decreased, unchanged or increased (PMR-AS < 10: decrease, PMR-AS > 17 increase to previous dosage, 10 ≤ PMR-AS ≤ 17: stable dose)
Medical resource evaluation | 36 weeks
  The cost of the utilization of Abatacept is evaluated
Following of the cumulative dosages of Glucocorticoids | 24 weeks
  The cumulative dosages of GCs is evaluated
The flare of the Polymyalgia Rheumatica | 36 weeks
  The flare of the Polymyalgia Rheumatica will be evaluate by the activity of Polymyalgia Rheumatica which is evaluated using the Polymyalgia Rheumatica Activity score ( (PMR-AS) which is not a scale but a score based on morning stiffness, ability to elevate the upper limbs, physician's global disease assessment and pain assessment measured by the patient using VAS, and the C-reactive protein (CRP) level. The PMR-AS is considered as relevant to define relapse and remission but also to decide if treatment have to be decreased, unchanged or increased (PMR-AS < 10: decrease, PMR-AS > 17 increase to previous dosage, 10 ≤ PMR-AS ≤ 17: stable dose).
Following of the medical exam using the ultrasound Scoring | 12 weeks
  The ultrasound scoring of synovitis and tenosynovitis is evaluated
Evaluation of FDG uptake using TEP-scanner in RegiOns of Interest | 12 weeks
  The FDG uptake is evalated with TEP-scanner using the FDG radiotracer
Following the proportion of patients relapse | 36 weeks
  The proportion of patients relapse or remission is evaluated with the Polymyalgia Rheumatica Activity score>17
Biological markers | 36 weeks
  The level of biological markers and cell subpopulations with the result of blood test is evaluated.
  The list of biological markers is (Interleukin, cytokines, immune cells)
Following of the quality of life | 36 weeks
  The Short Form 36 (SF36) is used to evaluate the quality of life. The SF36 scale includes 36 items divided into 8 dimensions (physical functioning, role limitations related to physical health, physical pain, general health, vitality [energy / fatigue].
Following of the quality of life | 36 weeks
  The scale EuroQol 5 dimensions (EDQ5) is used to evaluate the quality of life. The EQ-5D scale is a standardised measure of health status to provide a simple, generic measure of health for clinical and economic appraisal, whih is divided by the EQ-5D descriptive system (mobility, self care, usual activities, pain/discomfort, anxiety/depression) and the EQ Visual Analogue scale (EQ VAS). Each dimension has 5 levels (no problems, slight problems, moderate problems, severe problems, and extreme problems).
Following of the quality of life | 36 weeks
  The Hospital Anxiety and the Depression scale (HAD) is used to evaluate the quality of life.
  The HAD scale has 14 items rated from 0 to 3 with 7 questions relate to anxiety and 7 others to the depressive dimension.

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - CHRU de Brest, Brest
  - CH Le Mans, Le Mans
  - CH de Morlaix, Morlaix
  - CH St-Malo, St-Malo
  - CHU Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saraux A, Le Henaff C, Dernis E, Carvajal-Alegria G, Tison A, Quere B, Petit H, Felten R, Jousse-Joulin S, Guellec D, Marhadour T, Kervarrec P, Cornec D, Querellou S, Nowak E, Souki A, Devauchelle-Pensec V. Abatacept in early polymyalgia rheumatica (ALORS): a proof-of-concept, randomised, placebo-controlled, parallel-group trial. Lancet Rheumatol. 2023 Dec;5(12):e728-e735. doi: 10.1016/S2665-9913(23)00246-1. PMID 38251563
- [Derived] Allard B, Devauchelle-Pensec V, Saraux A, Nowak E, Tison A, Boukhlal S, Guellec D, Jousse-Joulin S, Cornec D, Marhadour T, Le Pennec R, Salaun PY, Querellou S. [18F]FDG PET/CT for therapeutic assessment of Abatacept in early-onset polymyalgia rheumatica. Eur J Nucl Med Mol Imaging. 2024 Apr;51(5):1297-1309. doi: 10.1007/s00259-023-06557-x. Epub 2023 Dec 14. PMID 38095675